CLINICAL TRIAL: NCT06230965
Title: Effect of Lung Protective Ventilation Strategy on Tumor Inflammatory Microenvironment and Its Associated Hematological Composite Index in Patients Undergoing Colorectal Cancer Surgery
Brief Title: Clinical Study of Lung Protective Ventilation Strategies and Tumor Microenvironment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yongtao Gao, Head of Anesthesiology, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: LPVS-MS2023025
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Tumor Microenvironment
Keywords: Lung protective ventilation strategies; Tumor microenvironment; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional ventilation strategy group (Other): The conventional ventilation strategy group used a conventional ventilation strategies: tidal volume（VT）=10-12 ml/kg, respiratory rate（f）=12 beats/minute, end-expiratory positive pressure（PEEP）= 0 cm H₂O, fraction of inspired oxygen = 0.5
  Interventions: Procedure: Lung protective ventilation strategy
- lung protective ventilation strategy group (Experimental): The lung protective ventilation strategy group used the lung protective ventilation strategies
  : tidal volume（VT）=6-8 ml/kg, f=12 breaths / minute,end-expiratory positive pressure（PEEP） = 6-8 cmH₂O, and fraction of inspired oxygen = 0.5 . After mechanical ventilation every 30 minutes (continuous positive airway pressure 30 cmH₂O for 30 seconds).
  Interventions: Procedure: Lung protective ventilation strategy

INTERVENTIONS:
Procedure: Lung protective ventilation strategy — They were divided into 2 groups: traditional ventilation strategy group (control group) and lung protective ventilation strategy group (experimental group), with 30 cases in each group. In the conventional ventilation strategy group, the conventional ventilation strategies were followed: tidal volume （VT）=10-12ml/kg, respiratory rate（f） =12 times/minute, PEEP=0 cmH₂O, fraction of inspired oxygen=0.5; Lung protective ventilation strategies were implemented in the Lung protective ventilation strategy group: VT=6-8ml/kg, f=12 times/min, PEEP=6-8 cm H₂O,fraction of inspired oxygen=0.5 Manual lung reexpansion was performed every 30 minutes after mechanical ventilation (continuous positive airway pressure of 30 cm H₂O for 30 seconds).
  Other Names: conventional ventilation strategy

SUMMARY:
This study will be conducted in the Affiliated Hospital of Nantong University. Sixty colorectal cancer(CRC) patients are randomized into traditional ventilation strategy group (control group) and lung protective ventilation strategy group (experimental group), there were 30 cases in each group. The control group adopted conventional ventilation strategy; the experimental group used lung protective ventilation strategy. 4ml of central venous blood was extracted at 3 time points within 24h, and relevant experimental indexes were determined. Observe the effect of lung protective ventilation strategy on the microenvironment of tumor inflammation and related hematological indexes in patients undergoing colorectal cancer surgery. Follow-up frailty score and quality of recovery score at 1,3,6, and 12 months after surgery (QoR-15 score scale).

DETAILED DESCRIPTION:
This study will be conducted in the Affiliated Hospital of Nantong University. Sixty CRC patients are randomized into traditional ventilation strategy group (control group) and lung protective ventilation strategy group (experimental group), there were 30 cases in each group. The control group adopted conventional ventilation strategies: tidal volume (VT)=10-12 ml/kg, respiratory rate ( f)=12 breaths / minute, positive end expiratory pressure（PEEP）=0 cmH₂O, fraction of inspired oxygen =0.5; the experimental group used lung protective ventilation strategies: tidal volume ( VT)=6-8 ml/kg, f=12 breaths / minute, positive end expiratory pressure (PEEP)=6-8 cmH₂O, fraction of inspired oxygen =0.5, mechanical ventilation every 30 minutes (continuous positive airway pressure 30 cmH₂O about 30 seconds). 4 ml of central venous blood was extracted at 3 time points within 24h, and relevant experimental indexes were determined. Observe the effect of lung protective ventilation strategy on the microenvironment of tumor inflammation and related hematological indexes NLDA, PDM, SII and PNI in patients undergoing colorectal cancer surgery. Follow-up frailty score and quality of recovery score at 1,3,6, and 12 months after surgery (QoR-15 score scale).

ELIGIBILITY:
Inclusion Criteria:

1. pathologic diagnosis of Colorectal Cancer
2. American society of Aneshesiologists（ASA）physical status classification system Grade Ⅱ-Ⅲ;
3. From 51-70 years old with no gender restrictions
4. Normal cardiopulmonary function before operation
5. Body Mass Index:18-30

Exclusion Criteria:

1. Preoperative anemia (hemoglobin<10g/dl)
2. Patients with preoperative mechanical ventilation;
3. A history of pulmonary infection and pulmonary tuberculosis within 1 month before surgery;
4. Preoperative blood oxygen saturation (SpO₂) was less than 90% (SpO₂<90%), or the oxygen partial pressure (PaO₂) was less than 90% (PaO₂<60 mmHg), or PaO₂/fraction of inspired oxygen（FiO₂）ratio<300 mmHg, or arterial blood carbon dioxide partial pressure (PaCO₂) was greater than 45 mmHg (PaCO₂>45 mmHg);
5. Patients who take immunosuppressants, neoadjuvant chemotherapy and radiotherapy before surgery;
6. Preoperative abnormal coagulation function.

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of tumor necrosis factor alpha (TNF-α)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of nucleartranscriptionfactorkappaB (NF-kB)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of interleukin-6 (IL-6)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of Tumor-associated macrophages (TAMs)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of vascular endothelial growth factor (VEGF)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of Janus Kinase 1 (JAK1)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of signal transducer and activator of transcription 3 (STAT3)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of Protooncogene tyrosine protein kinase (C-Src)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of matrix metalloproteinases 2 (MMP-2)
Microenvironment-related indicators of tumor inflammation | 10 minutes before anesthesia, 1 hour and 24 hours after the procedure
  Concentrations of matrix metalloproteinases 9 (MMP-9)

SECONDARY OUTCOMES:
Comprehensive blood index | 10 minutes before anesthesia and 24 hours after the procedure
  Values for NLDA (NLDA = neutrophil count/lymphocyte count × D-dimer count/albumin)
Comprehensive blood index | 10 minutes before anesthesia and 24 hours after the procedure
  Values for PDM (PDM = platelet× D-dimer count)
Comprehensive blood index | 10 minutes before anesthesia and 24 hours after the procedure
  Values for SII (SII= platelet× neutrophil / lymphocyte count)
Comprehensive blood index | 10 minutes before anesthesia and 24 hours after the procedure
  Values for PNI (PNI = albumin + 5 × lymphocytes)

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Gao, Master, Study Director — The Affiliated Hospital of Nantong University
Locations (1):
- The Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided